CLINICAL TRIAL: NCT00271466
Title: A Study to Assess the Safety, Dose Conversion and Titration of DURAGESIC® (Fentanyl Transdermal System) in Pediatric Subjects With Chronic Pain Requiring Opioid Therapy
Brief Title: A Study to Assess the Safety, Dose Conversion, and Dose Individualization of Duragesic® (Fentanyl Transdermal Patch) in the Treatment of Children With Chronic Pain Requiring Narcotic Pain Relief Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005977
Record Dates: First submitted 2005-12-30; First posted 2006-01-02 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Chronic Pain
Keywords: opioid; fentanyl; Duragesic; transdermal; chronic pain; morphine
MeSH Terms: conditions — Chronic Pain | interventions — Fentanyl

INTERVENTIONS:
Drug: DuragesicÂ® (fentanyl) Therapeutic Transdermal System (TTS)

SUMMARY:
The objective of this study is to assess the safety of treatment with Duragesic® (a transdermal patch delivering the narcotic pain-reliever fentanyl) in doses of 12.5, 25, 50, 75 and 100 micrograms/hour in pediatric subjects requiring narcotic pain relief therapy. Particular attention is paid to appropriate dose conversion to Duragesic® therapy from the subject's current narcotic pain relief therapy, and to the parameters for increasing the Duragesic® dose to achieve analgesic effectiveness. Pharmacokinetics (fentanyl levels in the bloodstream during treatment) will also be assessed.

DETAILED DESCRIPTION:
This is a single-arm, nonrandomized, open-label, multicenter trial designed to enroll a total of approximately 200 pediatric subjects with moderate to severe chronic pain due to malignant or nonmalignant disease. Subjects must have received opioids continuously for a minimum of 7 days prior to enrollment with a projected need for continuous opioids for at least the length of the primary treatment period. Subjects must also have received the equivalent of at least 30 mg of oral morphine on the day prior to enrollment. Subjects were enrolled into 3 age cohorts including 2 to <6 years, 6 to <12 years, and 12 to <16 years. The study consisted of a 15-day primary treatment period. After the 15-day primary treatment period, subjects may, at the investigator's discretion, continue long-term treatment with Duragesic® as long as medically appropriate. The objective of this study is to provide an evaluation of the safety of Duragesic® in pediatric subjects who require treatment with a potent opioid for the management of chronic pain. On Day 1, subjects are converted from oral or parenteral opioids to Duragesic® by calculating the previous 24-hour opioid analgesic requirement. This amount is then converted to the equi-analgesic oral morphine dose, and then used to determine the corresponding Duragesic® dose. Short-acting oral or parenteral opioids are used as rescue medication at any time during the study to treat breakthrough pain (pain not adequately controlled by Duragesic®). Following initiation of Duragesic® treatment using the recommended dose, subjects are titrated upwards (no more frequently than every 3 days after the initial dose) until analgesic effectiveness is attained. Titration is based on supplemental opioid consumption, such that the dose of Duragesic® is increased by 12.5 micrograms/hour for every 45 mg of oral morphine consumed on the 2nd or 3rd days following the last patch change, up to a maximum increase of 25 micrograms/hour at any one time. The primary endpoint of this trial is the determination of the safety profile of Duragesic® in the defined target population. Safety is assessed by monitoring adverse events, vital sign measurements, and through physical examination. In addition, respiratory rate and level of sedation are closely monitored during the first 72 hours. The assessment of clinical utility includes the parent's global assessment of pain control on Days 1 and 16, the pain level assessed by the parent and the patient twice daily, once in the morning and in the evening (or assessed by the parent only if the patient is younger than age 6), the pain level at the time rescue medication is given and one hour afterwards, the child's play performance, and a quality-of-life child health questionnaire (CHQ) used to measure the physical, psychosocial functioning and well being of children 5 years of age. During the primary treatment period, serum fentanyl concentrations are also measured. Sparse pharmacokinetic sampling is incorporated into the trial design to facilitate population pharmacokinetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from chronic pain of a well documented cause that requires continuous administration of opioids
* Received opioids continuously for a minimum of 7 days prior to enrollment with a projected need for continuous opioids for at least the length of the primary treatment period (15 days)
* Received the pain relief medication equivalent to at least 30 mg of oral morphine the day prior to enrollment
* Available for careful monitoring during the first 72 hours following administration of Duragesic®
* If female of child-bearing potential, must have a negative serum or urine pregnancy test within 1 week of enrollment

Exclusion Criteria:

* Patients with skin disease that precludes application of Duragesic® or which may affect the absorption of fentanyl
* Known sensitivity to fentanyl, other opioids, or adhesives
* Have a life expectancy less than the length of the primary treatment period (15 days)
* Have pain due to surgery, a clinically significant fever (i.e., above 38 C/100.4 F), a clinical condition that in the investigator's judgment prevents participation in the study (e.g., clinically significant liver or kidney dysfunction), or are currently being treated with ketoconazole, ritonavir or other disallowed concomitant therapy
* Female patients who are pregnant or breast feeding

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 199 (Actual)
Dates: Start 2000-02; Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events; Physical examination results and vital signs

SECONDARY OUTCOMES:
Parent's global assessment of pain control on Days 1 and 16; Pain level assessed once in the morning and in the evening; Pain level at the time rescue medication is given and one hour afterwards; Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Finkel JC, Finley A, Greco C, Weisman SJ, Zeltzer L. Transdermal fentanyl in the management of children with chronic severe pain: results from an international study. Cancer. 2005 Dec 15;104(12):2847-57. doi: 10.1002/cncr.21497. PMID 16284992
- See also: A study to assess the safety, dose conversion, and dose individualization of Duragesic® (fentanyl transdermal patch) in the treatment of children with chronic pain requiring narcotic pain relief therapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=698&filename=CR005977_CSR.pdf